CLINICAL TRIAL: NCT03672565
Title: Flexibly Dosed Intensive Exposure and Response Prevention as a Means to Maximize Outcomes for Youth With Obsessive Compulsive Disorder
Brief Title: SMART ERP for the Behavioral Treatment of Youth With Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Evelyn Stewart, MD, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H18-01654
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Exposure and Response prevention ERP; Cognitive-behavioural therapy; Pediatric OCD; Childhood-onset OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital setting (Active Comparator): ERPs may be conducted in various settings on hospital grounds (e.g., cafeteria, hallways) but will not be conducted off property.
  Interventions: Behavioral: Phase One: Standardized Brief Intensive ERP; Behavioral: Phase Two: Flexible Patient Driven Intensive ERP; Behavioral: Follow-Up Phase: Booster Calls
- Community setting (Active Comparator): Community ERP sessions will be conducted locations deemed most relevant to the child's symptom presentation such as in the home or at other community locations (e.g., church, downtown).
  Interventions: Behavioral: Phase One: Standardized Brief Intensive ERP; Behavioral: Phase Two: Flexible Patient Driven Intensive ERP; Behavioral: Follow-Up Phase: Booster Calls

INTERVENTIONS:
Behavioral: Phase One: Standardized Brief Intensive ERP — Participants will be randomized to receive ERP sessions at the hospital or at relevant community locations. In the introductory session, participants will be provided with psychoeducation about OCD and the treatment model, will develop a list of potential exposures, and will attempt initial exposure and response prevention (ERP) exercises. The session will end with an assignment of ERP homework. In the seven days following the introductory session, youth and parents will receive two 3-hour sessions, separated by a three day break. The sessions will begin with a brief review of homework completion and success. Following this, with parent observation, the clinician will guide the youth through escalating ERP exercises. The session will end with ERP homework planning. Other evidence-based treatment strategies (e.g., addressing motivation, discussing parental accommodations) may be implemented as deemed necessary by the clinician in order to encourage effective engagement in ERP exercises.
Behavioral: Phase Two: Flexible Patient Driven Intensive ERP — Families will have the opportunity to access up to four additional once/week 3-hour intensive ERP sessions.
  Three days prior to each additional ERP session (sessions 3-6), families will be prompted to fill out online forms and decide how to proceed with treatment for that week with the following options:
  * They may select that they would like to receive and complete the next ERP session, and up to four 3-hour ERP sessions during Phase Two. Completion of all four ERP session will automatically end Phase Two.
  * They may opt to delay receiving a treatment session by one week for any reason. Families will be allowed to take a week off up to two times during Phase Two. If both weeks off are utilized, at the next decision point families must either opt to complete an ERP Session or end their participation in Phase Two.
  * They may select to end their participation in Phase Two at any decision point and for any reason (e.g., don't perceive it as helpful, have improved substantially).
Behavioral: Follow-Up Phase: Booster Calls — Upon achieving remission at any remission assessment or completion of remission assessment five, youth will enter the follow-up phase. Youth will receive three weekly 30 minute post-treatment booster phone calls. Calls will focus on homework completion, ERP planning, and relapse prevention skills.

SUMMARY:
This randomized pilot study examines a graduated behavioral treatment approach for youth with obsessive compulsive disorder. Youth will be randomized to receive treatment in the community or at the hospital. In the first stage, youth receive an intro session and two 3-hour ERP sessions. Youth will be assessed for OCD recovery. Recovered youth enter follow-up. Still affected youth enter the second stage, where they will can select to receive up to four additional ERP sessions (one per week). In follow-up, youth will receive three 30 minute weekly calls and will be reassessed at 1- and 6-months following treatment.

DETAILED DESCRIPTION:
Obsessive compulsive disorder (OCD) is a highly debilitating psychiatric disorder that affects many youth. Despite strong empirical support that exposure and response prevention (ERP) is an efficacious and tolerable treatment of pediatric OCD including when presented in intensive formats, most individuals simply do not access or receive this treatment.

The dissemination of efficient interventions is of high public health priority, and graduated, or stepped care, models may be the answer. However, initial interventions within a graduated approach must be appropriate for the severity of the condition, given that unnecessary delays to an optimal dose may result in escalating burden on families and ultimately health services. Indeed, low intensity online CBT and self-help have so far had limited efficacy with less than one third of patients deemed responsive to treatment.

In contrast, brief intensive ERP is likely an efficient and effective alternative to flexibly dosing the level of intervention to the participant's needs. In fact, a recent pilot study (n = 10) providing two 3-hour ERP sessions to youth with OCD observed 60% post-treatment, and 70% 6-month follow-up, remission rates among participants. Extending on this study's findings, by utilizing more conservative remission criteria and providing access to additional doses of intensive ERP to youth not yet achieving remission, holds promise in identifying the level of services utilized by families to achieve meaningful treatment outcomes.

Above and beyond the use of a graduated dose model, many questions remain regarding optimal implementation methods for the behavioral treatment of pediatric OCD. In particular, the impact of treatment setting (i.e. community versus clinic) on response has not been systematically studied within this population. Given increased setting relevance and opportunity for in vivo learning, community exposures may be expected to be more effective; however, as they are associated with additional challenges (e.g., transportation time), their contribution to improvement needs to be directly verified and weighed against these costs.

Therefore, the present study seeks to determine the feasibility of implementing a sequential, multiple assignment, randomized trial (SMART) for the behavioral treatment of youth with OCD. The study focuses on evaluating the benefits from a minimum initial dose of intensive exposure and response prevention (ERP) as well as the demand for, and benefits from, additional ERP sessions by still-affected OCD families. In addition, via randomization, the study examines the influence of treatment setting (community vs hospital) on response. Primary outcomes include the impact of treatment on symptom severity and other relevant clinical outcomes (e.g., quality of life, youth- and family-functioning) as well as patient decisions/treatment utilization. Participant perspectives on study/treatment procedures (e.g., acceptability, optimal components) as well as cost-effectiveness (e.g., travel expenses, staff time, service utilization) will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 7 - 19 years
* Have a primary diagnosis of OCD
* Have a score of equal to, or greater than, 16 on the Children's Yale - Brown Obsessive Compulsive Scale
* Be, and have a parent/guardian, willing to participate in treatment
* Be stable on psychotropic medication as demonstrated by at least 10 weeks since first initiation of an serotonin reuptake inhibitor (SRI) and 4 weeks since initiation of any other psychotropic medications as well as 4 weeks since any dose adjustment of any psychotropic medications.
* Have sufficient English capabilities to complete questionnaires
* Live within the Greater Vancouver Area (within approximately 60 minutes drive of BC Children's Hospital)

Exclusion Criteria:

* Meet diagnostic criteria for bipolar disorder, psychosis, intellectual disability, substance dependence/abuse, or autism spectrum disorder (> level 1 impairment)
* Demonstrate alternate psychiatric symptoms of a more pressing nature than the OCD symptoms (e.g. suicidal intent in the context of comorbid depression)
* Youth or parents refusing to engage in treatment
* Initiation of an antidepressant within 10 weeks or an alternate psychotropic medication within 4 weeks or adjusted dosage within 4 weeks
* Family lives outside of the Greater Vancouver Area (longer than 60 minutes drive of BC Children's Hospital)

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Change in OCD symptom severity (i.e., percentage of youth achieving remission) following Treatment Phase One both within and between treatment settings (hospital vs. community) | Baseline Assessment (Week1/Day1), Post-treatment Assessment 1 (Week3/Day14)
  OCD symptom severity is measured with Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS), a clinician-rated scale of 10 items, each rated from 0 (no symptoms) to 4 (extreme symptoms), scores are summed to give a maximum score of 40. Higher scores indicate worse symptomatology. Youth will be identified as in remission if they are rated as having a total score of 11 (out of 40) or lower on the CY-BOCS at post-treatment assessment 1.
Change in OCD symptom severity between pre- and post-treatment for both treatment phases both within and between treatment settings | Phase 1: BA (Week1/Day1), PA1 (Week3/Day14) | Phase 2: TDP (weeks4-9/days18,25,32,39,46,53), PA2 (Week4-10/Day21,28,35,42,49,or60)
  OCD symptom severity is measured with Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS), a clinician-rated scale of 10 items, each rated from 0 (no symptoms) to 4 (extreme symptoms), scores are summed to give a maximum score of 40. Higher scores indicate worse symptomatology.
  Phase one pre- and post-treatment is assessed at Baseline assessment (BA) and PA1 while phase two pre- and post-treatment is assessed at Treatment Decision Point (TDP) and Post-treatment assessment 2 (PA2).
Number of sessions utilized by families used within treatment phase two both within and between treatment settings | TDP (Weeks4-9/Day18,25,32,39,46,or53)
  Following treatment phase one, families will decide between the following options at Treatment Decision Points (TDP):
  A) The family may select that they would like to receive and complete the next ERP session and can select to receive up to four additional 3-hour ERP sessions during Treatment Phase Two.
  B) The family may opt to delay receiving a treatment session by one week for any reason (e.g., prior engagement/holiday, additional time to evaluate symptoms). Families will be allowed to take a week off up to two times during Treatment Phase Two.
  C) The family may select to end their participation in Treatment Phase Two at any decision point and for any reason (e.g., don't perceive it as helpful, have improved substantially, have already utilized two weeks off and do not wish to have an additional session).

SECONDARY OUTCOMES:
Patient satisfaction and treatment tolerability | Treatment expectancy at Baseline Assessment; treatment perspectives at one-month follow-up following treatment completion
  Participant perspectives on study/treatment procedures (e.g., acceptability, optimal components) is measured with:
  * Treatment Expectancy Question (Clinician-, parent- and youth-rated forms)
  * Treatment Perspectives Form (Parent- and youth-rated)
Cost-effectiveness | After study completion
  Different aspects of cost-effectiveness will be examined (e.g., travel expenses, staff time, service utilization).
  A cost-utility analysis will be conducted to examine cost-benefit ratios between conditions and for the program as a whole.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn S. Stewart, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Selles RR, Naqqash Z, Best JR, Franco-Yamin D, Qiu ST, Ferreira JS, Deng X, Hannesdottir DK, Oberth C, Belschner L, Negreiros J, Farrell LJ, Stewart SE. Effects of Treatment Setting on Outcomes of Flexibly-Dosed Intensive Cognitive Behavioral Therapy for Pediatric OCD: A Randomized Controlled Pilot Trial. Front Psychiatry. 2021 May 17;12:669494. doi: 10.3389/fpsyt.2021.669494. eCollection 2021. PMID 34079488